CLINICAL TRIAL: NCT02701452
Title: Prevalence of Ovarian Hyperstimulation Syndrome in Patients Triggered by GnRH Agonist for Excessive Follicular Response After Ovarian Stimulation With a GnRH Antagonist
Brief Title: Ovarian Hyperstimulation Syndrome in Patients Triggered by GnRH Agonist for Excessive Follicular Response
Acronym: COAGO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014_08; 2015-A01291-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Hyperstimulation Syndrome; Hypercoagulability
Keywords: GnRH agonist triggering
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome; Thrombophilia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COAGO (Experimental): All patients undergoing antagonist protocol and at high risk of OHSS (estradiol level ≥ 3000 pg/mL and/or more than 20 follicles ≥ 11mm on the day of triggering) were triggered by GnRH agonist.
  Interventions: Other: COAGO

INTERVENTIONS:
Other: COAGO — blood samples for haemostasis and hormonal data

SUMMARY:
In the literature, the risk of moderate to severe OHSS is 3 to 6% and reaches 31% in high risk populations 9 days after oocyte triggering with hCG. Many studies report no or a markedly decreased risk of OHSS after triggering ovulation with a GnRH agonist. However, criteria to define OHSS are rarely explained and OHSS itself is not thoroughly asserted. It is well known that OHSS is associated with hypercoagulability. However, no study after triggering with a GnRH agonist assessed haemostasis in these high-risk patients with high circulating estradiol levels.

Study design, size, duration: In a French academic reproductive medicine centre, a systematic prospective observational follow-up of all patients triggered by GnRH agonist for excessive follicular response will be conducted. Participants/materials, setting, methods: All patients undergoing antagonist protocol and at high risk of OHSS (estradiol level ≥ 3000 pg/mL and/or more than 20 follicles ≥ 11mm on the day of triggering) will be triggered by GnRH agonist. No luteal phase support and a "freeze-all" strategy will be performed. On the day of oocyte retrieval (T0), at 48h (T1) and at day 7 (T2), OHSS and hypercoagulability will be systematically assessed. Haemostasis data will be compared to the initial status of each patient.

DETAILED DESCRIPTION:
Seventy-five patients will be required for this study.

ELIGIBILITY:
Inclusion Criteria:

* estradiol level ≥ 3000 pg/mL and/or more than 20 follicles ≥ 11mm on the day of triggering and antagonist protocol

Exclusion Criteria:

* agonist protocol no health assurance estradiol level < 3000 pg/mL and less than 20 follicles ≥ 11mm on the day of triggering

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with the presence of moderate to severe OHSS | The day of oocyte retrieval (Time 0).
  The OHSS defined by the classification of the "practice committee of the American Society for Reproductive Medicine" following biological, clinical and ultrasonographical criteria (composite):
  * Clinical: weight, waist circumference, dyspnea, EVA, diuresis
  * Organic: NFS, electrolytes, creatinine, urea, AST / ALT, albumin, serum protein
  * Ultrasound: ovarian size, quantification of ascites (Douglas, Morrison, parieto-colic gutters, vesico-uterine space).

SECONDARY OUTCOMES:
Dosage of Prothrombin time | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
Dosage of APTT | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
Dosage of fibrinogen | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
Dosage of von Willebrand factor antigen Antithrombin, | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
Dosage of DDimères | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
Dosage of oestradiol | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
  To evaluate its decrease.
Dosage of progesterone | The day of oocyte retrieval (Time 0), 2 days after (T1), 7 days after (T2), 6 weeks after (T3)
  To evaluate the quality of lutea and date of post punctures rules
Cumulative pregnancy rate after transfer of thawed embryos. | 2 months after the transfer of the last thawed embryo
Number of patients with the presence of moderate to severe OHSS | 2 days after (T1) and 7 days after (T2) the oocyte retrieval
  The OHSS defined by the classification of the "practice committee of the American Society for Reproductive Medicine" following biological, clinical and ultrasonographical criteria (composite):
  * Clinical: weight, waist circumference, dyspnea, EVA, diuresis
  * Organic: NFS, electrolytes, creatinine, urea, AST / ALT, albumin, serum protein
  * Ultrasound: ovarian size, quantification of ascites (Douglas, Morrison, parieto-colic gutters, vesico-uterine space).

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Catteau-Jonard, MD, PhD, Principal Investigator — University Hospital, Lille

IPD SHARING:
Plan to Share IPD: Undecided